CLINICAL TRIAL: NCT04099680
Title: Free Gingival Grafts (FGGs) in Mandibular Posterior Sites: A Randomized Clinical Trials of Wound Healing Following Different Recipient Bed Preparations
Brief Title: Free Gingival Grafts (FGGs) in Mandibular Posterior Sites
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fsafggrct2019; 2019H0350 (Other: Ohio State University IRB)
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-03

CONDITIONS: Lack of Keratinized Tissue
MeSH Terms: interventions — Bone Screws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Partial-thickness bed preparation (Active Comparator): Partial-thickness bed preparation for free gingival graft procedure.
  Interventions: Procedure: Partial thickness recipient bed; Procedure: Periosteal sutures; Procedure: Sling sutures
- Full-thickness bed preparation (Experimental): Full-thickness bed preparation with bone screw placement for anchoring the sutures.
  Interventions: Procedure: Full thickness recipient bed; Device: Bone screw (FDA approved bone screw); Procedure: Periosteal sutures; Procedure: Sling sutures around screws

INTERVENTIONS:
Procedure: Partial thickness recipient bed — Flap will be separated by sharp dissection and elevated toward apical direction, leaving the periosteum covering the bone, and the elevated pedicle flap will be incised and removed.
  Arms: Partial-thickness bed preparation
Procedure: Full thickness recipient bed — Full-thickness (mucoperiosteal) flap will be raised on the recipient bed to establish a denuded bone area. Two bone screws will be placed at the most apical border of the denuded bone.
  Arms: Full-thickness bed preparation
Device: Bone screw (FDA approved bone screw) — Two bone screws placed at the most apical border of the denuded bone after osteotomy.
  Arms: Full-thickness bed preparation
Procedure: Periosteal sutures — Interrupted periosteal sutures placed at the 4 corners of each graft, and mesial and distal surfaces to engage the graft at an equidistance from the graft corners.
Procedure: Sling sutures — Crossed sling sutures placed over the graft engaging the fixed crestal/lingual KT coronally and the periosteum apically.
  Arms: Partial-thickness bed preparation
Procedure: Sling sutures around screws — Crossed sling sutures placed over the graft engaging the fixed crestal/lingual KT coronally and each is apically looped around the corresponding apically positioned screw.
  Arms: Full-thickness bed preparation

SUMMARY:
In this proposed study a novel technique that utilizes bone screws as an anchorage device will be used to facilitate suturing and ensure graft tissue immobilization on full thickness recipient bed preparation sites. Currently, no information is available on free gingival graft treatment outcomes comparing full thickness recipient bed preparation, i.e., no periosteum remaining under the free gingival graft, with the aid of bone screws versus a conventional partial thickness recipient bed preparation with periosteum remaining under the graft. The purpose of the present study is to investigate the effect of these two different recipient bed preparations on soft tissue dimension change, graft and surgical wound healing, patient comfort, surgical complication frequency and operator satisfaction after free gingival graft to increase the width of keratinized gingival tissue in mandibular posterior sites. The purpose of the present study is to investigate the effect of these two different recipient bed preparations on soft tissue dimension change, graft and surgical wound healing, patient comfort, surgical complication frequency and operator satisfaction after free gingival graft procedure to increase the width of keratinized gingival tissue in mandibular posterior sites. The specific aims of this research study contain two aspects:

1. To compare the wound healing of a free gingival graft using either a partial thickness flap or full-thickness flap preparation with bone screws at the recipient site around mandibular posterior areas.
2. To assess patient comfort and surgeon satisfaction with a free gingival graft procedure using these two different recipient bed preparations.

DETAILED DESCRIPTION:
While the presence of a sufficient size of keratinized oral mucosa is favorable, the surgical procedure to increase the size is technically difficult. In the traditional way, preparation of the gum bed for a graft tissue is done with partial-thickness flap elevation, in which part of the mucosa and submucosa, but not the periosteum (dense fibrous membrane covering the surface of bones), are separated from underneath bone. In the traditional method of gum bed preparation, separation of the mucosa and submucosa from underneath periosteum and bone should be done with extremely caution to avoid damaging the periosteum. Therefore, the traditional method of gum bed preparation is not only time consuming but also problematic because of more bleeding when compared to full thickness flap elevation, in which the mucosa and submucosa together with the periosteum are separated from underneath bone. In order to stabilize gum graft on bone surface, a new technique is applied in this study by using two bone screws as anchorage to fastened the graft on the exposed bone through suturing. In the present study, we will compare patient quality of life, operator satisfaction, and differences in surgical wound healing between these two different bed preparations. The results of this study could help establish a more patient- and operator-friendly surgical protocol for the use of gum graft to increase the width of keratinized oral mucosa.

ELIGIBILITY:
A) Target population: Patients whether edentulous or dentate or treated with root-form dental implants, who need FGG on the buccal aspect of the mandibular posterior area.

Inclusion criteria <Demographic> Race: Any Non-smokers: No use of any tobacco or nicotine-replacement products for the least 5 years

<Medical history>

* Physically and mentally healthy with no contraindication for periodontal surgery
* American Society of Anesthesiologists: ASA-1 or ASA-2
* Clinical (Oral) conditions: Periodontally healthy patients with no contraindication for free gingival graft procedure (donor and recipient sites)

<Other>

* Patients who need free gingival graft in the mandibular posterior area.
* Patients who are able and willing to provide informed consent
* Patients who are able to receive surgery on Tuesday.

Exclusion criteria <Medical history>

* Smokers or users of nicotine replacement products
* Patients with any history of soft tissue surgery (grafting) in the area to be treated
* Patients with contraindication for periodontal soft tissue surgery, including an anatomical location of mental nerve that may restrict preparation of 10x10mm recipient bed
* Patients with contraindication, e.g., allergy, for any of the medications used in the study (benzocaine, lidocaine, chlorhexidine rinse, ibuprofen)
* Patients with inadequate donor site anatomy.
* Patients with uncontrolled diabetes (glycemic level > 110mg/l and HbA1c > 6%)
* Patients with drug or alcohol abuse
* Pregnant or lactating women
* Patients with a history of bisphosphonate therapy, radiotherapy in the head and neck region for malignancies, or chemotherapy for treatment of malignant tumors
* Other systemic conditions or medications affecting surgical or wound healing process and gingival tissues, such as cancer, HIV, metabolic bone diseases, phenytoin, cyclosporine, dihydropyridines, etc.

<Dental>

•Poor oral hygiene (PlI>2) 28

Subjects will be exited from the study immediately upon:

* Change of mind regarding participation
* Development of acute dental/oral conditions requiring treatment
* Development of a condition requiring treatment that conflicts with the exclusion criteria listed above
* Failure to comply with study instructions/requirements/appointments

B) Target population: Operators

Inclusion criteria

•2nd and 3rd year residents at Division of Periodontology, The Ohio State University, in good standing.

Exclusion criteria

•Residents who don't want to participate in the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Graft width, length and area | During the surgery, at the 1-, 2-, 4-, 8- week visits
  Graft length and width will be confirmed after harvest and remeasured in situ, using a digital caliper, after completion of the surgical procedure. Subsequently, graft length and width will be measured on clinical images obtained at the post-op visits. A mirror image photo of the grafted site will be taken with a single-lens reflex camera and the dimension will be measured and analyzed with Image J software. Size markers will be used to calibrate image magnification. Graft area will be calculated from the length and width measurements.

SECONDARY OUTCOMES:
Wound healing index | At the 3-day, 1-, 2-, 4-, 8- week visits
  Clinical photographs of the recipient sites will be taken at baseline, immediately after surgery, and at each follow-up visit, to record the appearance of the graft. A size marker will be used to standardize photos. Small size mirror will be placed with caution to avoid any disturbance of the surgical site, and mirror image photo will be taken. Wound healing index by Pippi et al. , which is the modified Wound Healing Index by Landry et al., is customized and used to evaluate the healing potential of the graft.
Graft thickness | During the surgery, at the 8-week visits
  Graft thickness will be measured in situ with digital caliper, and at the 8-week follow-up visit using an endodontic reamer, at five (5) predetermined points. A central point will be located at the geometric center of the graft, where the two diagonals of the square intersect. The other four points will each be located on the diagonal, at 3 mm from the corner of the graft. Pre-fabricated acrylic stent with holes for the measurements will be used to standardize measurement location. At 8 weeks, graft thickness measurements will be repeated following topical and local anesthesia using infiltration.
Graft mobility | At the end of surgery, at the 8-week visits
  At the end of the procedure, graft mobility will be assessed indirectly and graded. While exerting tension on the cheek/vestibule, graft will be observed for mobility. Mobility will be graded indirectly, by exerting tension on the cheek/vestibule, and directly, by applying gentle force on the graft using a periodontal probe, in a manner similar to the functional approach used to locate the mucogingival junction.
Biochemical wound assessment | At the 3-day, 1-, 2- week visits
  Wound fluid will be collected from the transplanted graft site. Paper strips will be left in place for 30 sec and then immediately transferred to a micro-moisture meter to determine the volume of collected fluid. Following volume measurement, paper strips will be immediately placed into a vial, on ice; fluid collection will be repeated after 5 minutes. Then the vial with the 4 paper strips will be transferred to a -80˚C freezer until further analysis. Expression of angiogenesis biomarkers will be quantified with the use of a human angiogenesis custom array kit according to the manufacturer's protocol.
Surgical time | During the surgery
  Length of surgery will be measured at the time the operator starts the first incision in the recipient bed and stopped when the last suture placement is placed. Bed preparation and graft placement will be independently timed to compare between procedures and with operator's opinion.
Pain assessment. | At the 3-day, 1-, 2-, 4-, 8- week visits
  A visual analogue scale (VAS) will be used to measure daily pain intensity at each postoperative week. The self-reported degree of pain will be scored, with 0 defined as the absence of pain and 10 as the maximum tolerable level of pain. The intake of NSAIDs will be also recorded. .
OHIP-14 | Right before the surgery and at the 3-day, 1-, 2-, 4-, 8- week visits
  The oral health-related quality of life will be assessed by the Oral Health Impact Profile scale (OHIP-14). Participants will be asked how frequently they had experienced the impact on each category in OHIP-14 with a 5-point scale (from 0 to 4). The total score of OHIP-14 will be calculated by adding the sum of each category from 14 questions (total score ranges from 0 to 56 points). Higher scores imply a poorer oral health quality of life, whereas lower scores indicate a better one.
Operator-centered outcomes | Immediately after the surgery, 2-week post-op visit and when an operator has conducted all allocated cases
  Immediately after the surgery, operators will receive custom questionnaire to assess the difficulty of the surgery. Each step of the surgery will be categorized and will be marked with 10-point scale (from 0 to 10) based on the surgical difficulty and time management.
  After completion of the 2-week post-op visit, operators will be asked to assess difficulty of screw removal (test group only).
  Also, after each enrolled operator has conducted all allocated cases (2 cases of full-thickness flap group and 2 cases of partial-thickness flap group, possibly up to 1 year.), including all 2-week post-op visits, he/she will be asked to report their preference of procedure (control or test)

CONTACTS AND LOCATIONS:
Overall Officials: Tatakis Dimitris, DDS, PhD, Study Director — The Ohio State University Graduate Periodontics Program Director
Locations (1):
- The Ohio State University College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoma DS, Buranawat B, Hammerle CH, Held U, Jung RE. Efficacy of soft tissue augmentation around dental implants and in partially edentulous areas: a systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S77-91. doi: 10.1111/jcpe.12220. PMID 24641003
- [Background] Nabers JM. Free gingival grafts. Periodontics. 1966 Sep-Oct;4(5):243-5. No abstract available. PMID 5223124
- [Background] Sullivan HC, Atkins JH. Free autogenous gingival grafts. I. Principles of successful grafting. Periodontics. 1968 Jun;6(3):121-9. No abstract available. PMID 5240496
- [Background] Sullivan HC, Atkins JH. Free autogenous gingival grafts. 3. Utilization of grafts in the treatment of gingival recession. Periodontics. 1968 Aug;6(4):152-60. No abstract available. PMID 5243142
- [Background] Dorfman HS, Kennedy JE, Bird WC. Longitudinal evaluation of free autogenous gingival grafts. J Clin Periodontol. 1980 Aug;7(4):316-24. doi: 10.1111/j.1600-051x.1980.tb01974.x. PMID 6936409
- [Background] Dorfman HS, Kennedy JE, Bird WC. Longitudinal evaluation of free autogenous gingival grafts. A four year report. J Periodontol. 1982 Jun;53(6):349-52. doi: 10.1902/jop.1982.53.6.349. PMID 7050339
- [Background] Kennedy JE, Bird WC, Palcanis KG, Dorfman HS. A longitudinal evaluation of varying widths of attached gingiva. J Clin Periodontol. 1985 Sep;12(8):667-75. doi: 10.1111/j.1600-051x.1985.tb00938.x. PMID 3902907
- [Background] Lang NP, Loe H. The relationship between the width of keratinized gingiva and gingival health. J Periodontol. 1972 Oct;43(10):623-7. doi: 10.1902/jop.1972.43.10.623. No abstract available. PMID 4507712
- [Background] Miyasato M, Crigger M, Egelberg J. Gingival condition in areas of minimal and appreciable width of keratinized gingiva. J Clin Periodontol. 1977 Aug;4(3):200-9. doi: 10.1111/j.1600-051x.1977.tb02273.x. PMID 330574
- [Background] Scheyer ET, Sanz M, Dibart S, Greenwell H, John V, Kim DM, Langer L, Neiva R, Rasperini G. Periodontal soft tissue non-root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S73-6. doi: 10.1902/jop.2015.140377. PMID 25644301
- [Background] Gobbato L, Avila-Ortiz G, Sohrabi K, Wang CW, Karimbux N. The effect of keratinized mucosa width on peri-implant health: a systematic review. Int J Oral Maxillofac Implants. 2013 Nov-Dec;28(6):1536-45. doi: 10.11607/jomi.3244. PMID 24278922
- [Background] Brito C, Tenenbaum HC, Wong BK, Schmitt C, Nogueira-Filho G. Is keratinized mucosa indispensable to maintain peri-implant health? A systematic review of the literature. J Biomed Mater Res B Appl Biomater. 2014 Apr;102(3):643-50. doi: 10.1002/jbm.b.33042. Epub 2013 Oct 7. PMID 24124021
- [Background] Wennstrom JL, Bengazi F, Lekholm U. The influence of the masticatory mucosa on the peri-implant soft tissue condition. Clin Oral Implants Res. 1994 Mar;5(1):1-8. doi: 10.1034/j.1600-0501.1994.050101.x. PMID 8038340
- [Background] Adibrad M, Shahabuei M, Sahabi M. Significance of the width of keratinized mucosa on the health status of the supporting tissue around implants supporting overdentures. J Oral Implantol. 2009;35(5):232-7. doi: 10.1563/AAID-JOI-D-09-00035.1. PMID 19882819
- [Background] Martin W, Lewis E, Nicol A. Local risk factors for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:28-38. PMID 19885433
- [Background] Schrott AR, Jimenez M, Hwang JW, Fiorellini J, Weber HP. Five-year evaluation of the influence of keratinized mucosa on peri-implant soft-tissue health and stability around implants supporting full-arch mandibular fixed prostheses. Clin Oral Implants Res. 2009 Oct;20(10):1170-7. doi: 10.1111/j.1600-0501.2009.01795.x. Epub 2009 Aug 30. PMID 19719741
- [Background] Abrahamsson I, Berglundh T, Wennstrom J, Lindhe J. The peri-implant hard and soft tissues at different implant systems. A comparative study in the dog. Clin Oral Implants Res. 1996 Sep;7(3):212-9. doi: 10.1034/j.1600-0501.1996.070303.x. PMID 9151585
- [Background] Jansen JA, de Wijn JR, Wolters-Lutgerhorst JM, van Mullem PJ. Ultrastructural study of epithelial cell attachment to implant materials. J Dent Res. 1985 Jun;64(6):891-6. doi: 10.1177/00220345850640060601. PMID 2987325
- [Background] Ericsson I, Berglundh T, Marinello C, Liljenberg B, Lindhe J. Long-standing plaque and gingivitis at implants and teeth in the dog. Clin Oral Implants Res. 1992 Sep;3(3):99-103. doi: 10.1034/j.1600-0501.1992.030301.x. PMID 1290796
- [Background] Lin GH, Chan HL, Wang HL. The significance of keratinized mucosa on implant health: a systematic review. J Periodontol. 2013 Dec;84(12):1755-67. doi: 10.1902/jop.2013.120688. Epub 2013 Mar 1. PMID 23451989
- [Background] Dordick B, Coslet JG, Seibert JS. Clinical evaluation of free autogenous gengival grafts placed on alveolar bone. Part I. Clinical predictability. J Periodontol. 1976 Oct;47(10):559-67. doi: 10.1902/jop.1976.47.10.559. PMID 1067398
- [Background] Caffesse RG, Burgett FG, Nasjleti CE, Castelli WA. Healing of free gingival grafts with and without periosteum. Part I. Histologic evaluation. J Periodontol. 1979 Nov;50(11):586-94. doi: 10.1902/jop.1979.50.11.586. No abstract available. PMID 115984
- [Background] James WC, McFall WT Jr. Placement of free gingival grafts on denuded alveolar bone. Part I: clinical evaluations. J Periodontol. 1978 Jun;49(6):283-90. doi: 10.1902/jop.1978.49.6.283. PMID 279658
- [Background] Nobuto T, Imai H, Yamaoka A. Microvascularization of the free gingival autograft. J Periodontol. 1988 Oct;59(10):639-46. doi: 10.1902/jop.1988.59.10.639. PMID 3183914
- [Background] Yanagihara K. [Experimental studies on morphological changes of microvascular architecture following the free gingival autograft on denuded alveolar bone]. Nihon Shishubyo Gakkai Kaishi. 1990 Mar;32(1):45-70. doi: 10.2329/perio.32.45. Japanese. PMID 1724261
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Egbewale BE. Random allocation in controlled clinical trials: a review. J Pharm Pharm Sci. 2014;17(2):248-53. doi: 10.18433/j3sw36. PMID 24934553
- [Background] Pippi R, Santoro M, Cafolla A. The effectiveness of a new method using an extra-alveolar hemostatic agent after dental extractions in older patients on oral anticoagulation treatment: an intrapatient study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2015 Jul;120(1):15-21. doi: 10.1016/j.oooo.2015.02.482. Epub 2015 Mar 2. PMID 25817129
- [Background] Guglielmoni P, Promsudthi A, Tatakis DN, Trombelli L. Intra- and inter-examiner reproducibility in keratinized tissue width assessment with 3 methods for mucogingival junction determination. J Periodontol. 2001 Feb;72(2):134-9. doi: 10.1902/jop.2001.72.2.134. PMID 11288784
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Landry R, Turnbull R, Rochette C. Effectiveness of benzydamyne HCl in the treatment of periodontal post-surgical patients. Res Clin Forums. 1988;10:105-18.
- [Result] Silva CO, Ribeiro Edel P, Sallum AW, Tatakis DN. Free gingival grafts: graft shrinkage and donor-site healing in smokers and non-smokers. J Periodontol. 2010 May;81(5):692-701. doi: 10.1902/jop.2010.090381. PMID 20429648